CLINICAL TRIAL: NCT01419327
Title: Special Drug Use Investigation of Fosrenol (Long-term Investigation for Patients With Hemodialysis)
Brief Title: Fosrenol Post-marketing Surveillance for Hemodialysis in Japan
Acronym: FOSRENOL-HD
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15077
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Hyperphosphatemia
Keywords: Fosrenol; Hyperphosphatemia; Hemodialysis
MeSH Terms: conditions — Hyperphosphatemia | interventions — lanthanum carbonate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Drug (incl. Placebo)
  Interventions: Drug: Lanthanum Carbonate (Fosrenol, BAY77-1931) - chewable tablet

INTERVENTIONS:
Drug: Lanthanum Carbonate (Fosrenol, BAY77-1931) - chewable tablet — Patients in hemodialysis who have received Fosrenol for hyperphosphatemia.

SUMMARY:
This study is a regulatory post marketing surveillance in Japan, and it is a local prospective and observational study of patients in hemodialysis who received Fosrenol for hyperphosphatemia. The objective of this study is to assess safety and efficacy of using Fosrenol in clinical practice. A total 3,000 patients will be recruited and followed 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hemodialysis who received Fosrenol for hyperphosphatemia

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is patients who have received a prescription of Fosrenol on the basis of the decision of the physician. The study is expected to collect data of 3,000 patients in about 300 practices in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 3267 (Actual)
Dates: Start 2009-03-23 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions in subjects who received Fosrenol | After Fosrenol administration, up to 8 years

SECONDARY OUTCOMES:
Timing of onset of common ADRs related to the priority survey items | After Fosrenol administration, up to 8 years
  The items are
  * Gastrointestinal symptoms
  * Secondary hyperparathyroidism
  * Hypocalcaemia and decreased blood calcium
Effect on bones: Alkaline phosphatase over time | After Fosrenol administration, up to 8 years
Effect on bones: Change in bone density | After Fosrenol administration, up to 8 years
Cardiothoracic ratio over time | After Fosrenol administration, up to 8 years
PWV and ABI over time | After Fosrenol administration, up to 8 years
Serum P, albumin-corrected serum Ca and serum intact PTH, and Ca-P product over time | After Fosrenol administration, up to 8 years
Percentage of patients achieving the serum P control goal | After Fosrenol administration, up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/